CLINICAL TRIAL: NCT03145974
Title: Prevalence and Outcome of Acute Hypoxemic Respiratory Failure (PANDORA Study)
Brief Title: Prevalence and Outcome of Acute Hypoxemic Respiratory Failure
Acronym: PANDORA
Status: Completed | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Collaborators: Asociación Científica Pulmón y Ventilación Mecánica (Other); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Principal Investigator, Jesus Villar, Clinical scientist, Dr. Negrin University Hospital
Other Study IDs: ACPVM170501
Record Dates: First submitted 2017-04-19; First posted 2017-05-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2018-07

CONDITIONS: Acute Respiratory Insufficiency
Keywords: respiratory failure; mechanical ventilation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypoxemic Acute Respiratory Failure: Consecutive intubated patients receiving invasive mechanical ventilation, with a PaO2/FiO2 ≤300 mmHg under a PEEP of 5 cmH2O or more, and with a FiO2 of 0.3 or more.
  Interventions: Device: mechanical ventilation

INTERVENTIONS:
Device: mechanical ventilation — ventilatory support

SUMMARY:
This study is an extension of the Spanish Initiative for Epidemiology, Stratification and Therapies of Acute respiratory failure (SIESTA) Network.

The present study is aimed to establish the epidemiological characteristics and clinical outcomes of mechanically ventilated patients with acute hypoxemic respiratory failure [defined as a PaO2/FiO2 ≤300 mmHg on positive end-expiratory pressure (PEEP) of 5 cmH2O or more, and FiO2 of 0.3 or more] admitted in a network of Spanish hospitals.

DETAILED DESCRIPTION:
The present study is aimed to establish the epidemiological characteristics and clinical outcomes of adult mechanically ventilated patients with acute hypoxemic respiratory failure [defined as a PaO2/FiO2 ≤300 mmHg on positive end-expiratory pressure (PEEP) of 5 cmH2O or more and FiO2 of 0.3 or more] admitted in a network of Spanish hospitals. Although there are few previous published observational studies examining the incidence and mortality of patients with acute respiratory failure and ARDS, there are no studies specifically assessing the epidemiological characteristics, patterns of ventilation and clinical outcomes in patients with acute hypoxemic respiratory failure in the current era of lung protective ventilation.

Since the study is prospective, with consecutive collection of clinically relevant data from patients and with the participation of several ICUs from different geographical regions of Spain, the findings would be highly generalizable. The study is aimed to improve the knowledge on the epidemiology and outcome of ventilated patients, to identify the percentage of patients developing ARDS under the current definition, to validate a bedside scoring system developed by us for stratification of lung severity, and to examine the prognosis of hypoxemic respiratory failure, and risk factors associated with fatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18-year old.
* Endotracheal intubation and mechanical ventilation, independent of whether the need for ventilatory support is shorter or longer than 24 hours. Only patients receiving invasive mechanical ventilation can be included, although patients could have been on non-invasive ventilation before intubation.
* PaO2/FiO2 ≤300 mmHg on invasive mechanical ventilation with a PEEP of 5 cmH2O or more, and with a FiO2 of 0.3 or more.

Exclusion Criteria:

* No patients should be excluded (if they meet all the inclusion criteria), regardless of the underlying disease, estimated life expectancy, or duration of invasive mechanical ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted to participating ICUs will be screened daily. Only patients meeting inclusion criteria for acute hypoxemic respiratory failure (as defined above) will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of hypoxemic acute respiratory failure | 6 months
  The investigators will calculate the prevalence in relation to: (i) total number of ICU admissions during the study period in all participating centers; (ii) total number of mechanically ventilated patients during the study period in all participating centers, and (iii) per ICU bed available in the participating centers over the study period.

SECONDARY OUTCOMES:
death in the ICU | Intensive care unit stay [up to 60 days]
  outcome at the time of discharge from ICU
death in the hospital | Hospital stay [Maximum 6 months]
  outcome before discharge to home (overall and in each category of acute hypoxemic respiratory failure).

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Villar, MD, PhD, Principal Investigator — Hospital Dr. Negrin, Las Palmas de Gran Canaria, Spain
Locations (24):
- Spain (24):
  - Complejo Hospitalario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitario Mutua de Terrasa, Terrassa, Barcelona
  - Hospital La Mancha Centro, Alcázar de San Juan, Ciudad Real
  - Hospital El Bierzo, Ponferrada, León
  - Hospital Universitario NS de Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital NS del Prado, Talavera de la Reina, Toledo
  - Hospital Universitario de La Coruña, A Coruña
  - Complejo Hospitalario de Albacete, Albacete
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital Virgen de La Luz, Cuenca
  - Complejo Hospitalario Universitario de León, León
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen de Arrixaca, Murcia
  - Hospital General de Segovia, Segovia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Hospital Universitario Rio Hortega - Anesthesia, Valladolid
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Virgen de la Concha, Zamora

IPD SHARING:
Plan to Share IPD: No
Patients' data will be anonymized and recorded in a case report form (CRF) specifically designed for this study. Data will be presented globally at the end of the study

REFERENCES:
- [Derived] Villar J, Gonzalez-Martin JM, Ambros A, Mosteiro F, Martinez D, Fernandez L, Soler JA, Parra L, Solano R, Soro M, Del Campo R, Gonzalez-Luengo RI, Civantos B, Montiel R, Pita-Garcia L, Vidal A, Anon JM, Ferrando C, Diaz-Dominguez FJ, Mora-Ordonez JM, Fernandez MM, Fernandez C, Fernandez RL, Rodriguez-Suarez P, Steyerberg EW, Kacmarek RM; Spanish Initiative for Epidemiology, Stratification and Therapies of ARDS (SIESTA) Network. Stratification for Identification of Prognostic Categories In the Acute RESpiratory Distress Syndrome (SPIRES) Score. Crit Care Med. 2021 Oct 1;49(10):e920-e930. doi: 10.1097/CCM.0000000000005142. PMID 34259448